CLINICAL TRIAL: NCT02789332
Title: A Randomized Phase II Trial to Assess the Efficacy of Paclitaxel and Olaparib in Comparison to Paclitaxel / Carboplatin Followed by Epirubicin/Cyclophosphamide as Neoadjuvant Chemotherapy in Patients With HER2-negative Early Breast Cancer and Homologous Recombination Deficiency (HRD Patients With Deleterious BRCA1/2 Tumor or Germline Mutation and/or HRD Score High)
Brief Title: Assessing the Efficacy of Paclitaxel and Olaparib in Comparison to Paclitaxel / Carboplatin Followed by Epirubicin/Cyclophosphamide as Neoadjuvant Chemotherapy in Patients With HER2-negative Early Breast Cancer and Homologous Recombination Deficiency
Acronym: GeparOla
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG90
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Triple Negative Breast Neoplasms; HRpos Breast Neoplasms; BRCA 1 /2 and / or HRD
Keywords: carboplatin; olaparib; pCR; neoadjuvant; triple-negative; hormonreceptor-positive; BRCA1/2; HRD, homologous recominant deficient; breast cancer; genetic testing (somatic and germline mutations)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Kenny-Caffey syndrome, Type 1 | interventions — Epirubicin; Cyclophosphamide; Vernalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel with Carboplatin (PwCb) (Active Comparator): paclitaxel 80 mg/m² iv weekly in combination with carboplatin AUC 2 iv weekly for 12 weeks (37 patients) followed by 4 cycles of epirubicin 90 mg/m² and cyclophosphamide 600 mg/m² (EC) either every 3 or every 2 weeks followed by surgery.
  Interventions: Drug: PwCb; Drug: EC; Procedure: Surgery after neoadjuvant Therapy; Other: Stratification
- Paclitaxel with Olaparib (PwO) (Experimental): paclitaxel 80 mg/m² iv weekly in combination with olaparib tablets 100 mg twice daily for 12 weeks (65 patients)
  followed by 4 cycles of epirubicin 90 mg/m² and cyclophosphamide 600 mg/m² (EC) either every 3 or every 2 weeks followed by surgery.
  Interventions: Drug: PwO; Drug: EC; Procedure: Surgery after neoadjuvant Therapy; Other: Stratification

INTERVENTIONS:
Drug: PwO — paclitaxel 80 mg/m² iv weekly in combination with olaparib tablets 100 mg twice daily for 12 weeks (PwO) (65 patients)
  Other Names: Paclitaxel Olaparib over 12 weeks
  Arms: Paclitaxel with Olaparib (PwO)
Drug: PwCb — paclitaxel 80 mg/m² iv weekly in combination with carboplatin AUC 2 iv weekly for 12 weeks (PwCb) (37 patients)
  Other Names: Paclitaxel Carboplatin over 12 weeks, Control arm currently considered standard of care regimen
  Arms: Paclitaxel with Carboplatin (PwCb)
Drug: EC — both Arms followed by 4 cycles of epirubicin 90 mg/m² and cyclophosphamide 600 mg/m² (EC) either every 3 or every 2 weeks followed by surgery.
  Other Names: Epirubicin 90 mg/m² and Cyclophosphamide 600 mg/m² (EC) either every 3 or every 2 weeks
Procedure: Surgery after neoadjuvant Therapy — In both study arms, treatment will be given until surgery, disease progression, unacceptable toxicity, or withdrawal of consent of the patients.
Other: Stratification — Hormone-receptor status (HR+ vs HR-) Age < 40 years vs >= 40 years
  Other Names: Randomization will be performed using Pocock minimization method, stratified for the following criteria:

SUMMARY:
This is a multicenter, prospective, randomized, open-label phase II study evaluating the efficacy and safety of PO→EC as neoadjuvant treatment of operable and locally advanced breast cancer in patients with HR deficiency. Patients will be randomized to receive

* paclitaxel 80 mg/m² iv weekly in combination with olaparib tablets 100 mg (4X25mg) twice daily for 12 weeks (65 patients) or
* paclitaxel 80 mg/m² iv weekly in combination with carboplatin AUC 2 iv weekly for 12 weeks (37 patients) both followed by 4 cycles of epirubicin 90 mg/m² and cyclophosphamide 600 mg/m² (EC) either every 3 or every 2 weeks followed by surgery.

The control arm was chosen to allow direct comparison with one of the currently considered standard of care regimen.

DETAILED DESCRIPTION:
The efficacy of olaparib in germline HRD score high with or without BRCA 1/2 mutation carriers with breast cancer is not well described

* The efficacy and safety of olaparib included in a standard of care regimen like paclitaxel weekly followed by epirubicin and cyclophosphamide (Pw-->EC) is unknown
* Carboplatin increased the pCR rate in patients with triple-negative breast cancer (TNBC) in two randomized phase II neoadjuvant studies when added to an anthracycline, cyclophosphamide and paclitaxel (GeparSixto, CALBG 40603). pCR rates were even higher in patients with germline BRCA 1 or 2 mutations (ypT0/is ypN0 65%) and with HRD score high (ypT0/is ypN0 63%).
* The TNT study showed a doubling in response rate for patients receiving carboplatin vs docetaxel in patients with germline BRCA 1 or 2 mutations.
* There is a high correlation between tumor and germline BRCA 1/2 mutations.
* Data from Geparsixto study showed that triple negative breast patients have an HR deficiency in about 70% (67% have a high HRD and 30% have a tBRCA mutation)
* About 5% of tBRCA patients have a low HRD score
* gBRCA2 patients are older when diagnosed and are more likely to have an HRpos tumor.
* The GeparOLA study aims to support the decision for a phase III study exploring the addition of olaparib to a Pw-->EC schedule by providing an estimate on the pCR rate in the targeted population but also by providing estimate comparison to paclitaxel and carboplatin followed by epirubicin and cyclophosphamide (PCb-->EC) as carboplatin is more and more considered a standard option of care in HR deficient patients (tBRCA 1/2 mutations and/or HRD score high).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study specific procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Complete baseline documentation must be sent to GBG Forschungs GmbH.
3. Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
4. Centrally confirmed negative HER2-status. Centrally confirmed estrogen and progesterone receptor, and Ki-67 status detected on core biopsy. ER/PR positive is defined as ≥1% stained cells and HER2-positive is defined as IHC 3+ or in-situ hybridisation (ISH) ratio ≥2.0. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy has therefore to be sent to the Dept. of Pathology at the Charité, Berlin prior to randomization.
5. Centrally confirmed tumor Homologous Recombinant Deficiency score (tBRCA positive/mutated and/or HRD high). Patients with known gBRCA and/or tBRCA status can be enrolled prior to the central test results available.
6. Tumor lesion in the breast with a palpable size of > 2 cm or a sonographical size of >1 cm in maximum diameter. If the tumor is not detectable with sonography mammography assessment can be considered. The lesion has to be measurable in two dimensions, preferably by sonography. In case of inflammatory disease, the extent of inflammation can be used as measurable lesion.
7. Patients must be in the following stages of disease:

   * cT2 - cT4a-d or
   * cT1c and cN+ or cT1c and pNSLN+ or
   * cT1c and ER-neg and PR-neg or
   * cT1c and Ki67>20% In patients with multifocal or multicentric breast cancer, the largest lesion should be measured and at least one lesion has to meet the above criteria
8. Age > 18 years.
9. Karnofsky Performance status index ≥ 80%.
10. Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results must be above the normal limit of the institution.
11. Laboratory requirements:

    Hematology
    * Absolute neutrophil count (ANC) ≥2.0 x 109 / L and
    * Platelets ≥100 x 109 / L and
    * Hemoglobin ≥10 g/dL (≥ 6.2 mmol/L) Hepatic function
    * Total bilirubin ≥1.5x UNL and
    * ASAT (SGOT) and ALAT (SGPT) ≥1.5x UNL and
    * Alkaline phosphatase ≥2.5x UNL.
12. Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential.
13. Complete staging work-up within 3 months prior to randomization. All patients must have bilateral mammography, breast ultrasound (≥21 days, and in no case exceed 6 weeks prior to randomization) (Note MRI/ CT scan may be used as an alternative imaging technique). In case of high risk according to guidelines: chest X-ray (PA and lateral) or as an alternative breast MRI/CT, abdominal ultrasound or CT scan or MRI, and bone scan in case of high risk for primary metastasis according to guidelines. In case of positive bone scan, bone X-ray or CT scan is mandatory. Other tests may be performed as clinically indicated.
14. Male or female patients
15. Patients must be available and compliant for central diagnostics, treatment and follow-up.

Exclusion Criteria:

1. Prior chemotherapy for any malignancy within 5 years.
2. Prior radiation therapy for breast cancer within 5 years.
3. Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization) during study treatment.
4. Inadequate general condition (not fit for anthracycline-taxane-targeted agents-based chemotherapy).
5. Previous malignant disease without being disease-free for less than 5 years (except CIS of the cervix and non-melanomatous skin cancer).
6. Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >140 / 90 mm Hg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
7. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
8. Patients currently in an institution by order of jurisdictional or governmental grounds.
9. Currently active infection.
10. Definite contraindications for the use of corticosteroids.
11. Known hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol.
12. Concurrent treatment with:

    * chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (10 mg or less methylprednisolone or equivalent).
    * sex hormones. Prior treatment must be stopped before study entry.
    * other experimental drugs or any other anti-cancer therapy.
13. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
14. Prior use of a PARP-Inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
response by pCR =ypT0/is ypN0 | 24 weeks
  Assess the efficacy of olaparib in HER2-negative early Breast Cancer and HRD (BRCA 1/2 mutations and/or HRD positive). Pathological complete response of breast and lymph nodes (ypT0/is ypN0) defined as no microscopic evidence of residual invasive viable tumor cells in all resected specimens of the breast and axilla.
  Pathological response will be assessed considering all removed breast and lymphatic tissues from all surgeries.

SECONDARY OUTCOMES:
response by pCR =ypT0/is ypN0 | 12 weeks
  To assess the pCR rates of patients receiving PO→EC and the pCR rates of patients receiving paclitaxel and carboplatin followed by EC (PCb→EC)
response by pCR =ypT0/is ypN0 in stratified subgroups | 24 weeks
  To assess the pCR rates (ypT0/is, ypN0) in the stratified subgroups
response by pCR according to other definitions | 24 weeks
  To determine other pCR rates (ypT0 ypN0; ypT0 ypN0/+; ypT0/is ypN0/+; ypT(any) ypN0) of patients receiving PO→EC and to compare them with the pCR rates of patients receiving PCb→EC.
response by pCR in HRD high versus tBRCA | 24 weeks
  To assess the pCR rate in HRD high with vs without tBRCA mutation
Response rate by sono and/or mammo | 12 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) with PO→EC and to compare it with PCb→EC. Clinical (c) and imaging (i) response will be assessed after EC and before surgery by physical examination and imaging tests. Sonography is the preferred examination, however, if sonography appears not to provide valid results or is not performed, other imaging tests will be considered.
Response rate by sono and/or mammo | 24 weeks
  To determine the response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) with PO→EC and to compare it with PCb→EC. Clinical (c) and imaging (i) response will be assessed after EC and before surgery by physical examination and imaging tests. Sonography is the preferred examination, however, if sonography appears not to provide valid results or is not performed, other imaging tests will be considered.
Breast Conservation rate | 24 weeks
  To determine the breast conservation rate with PO→EC and to compare it with PCb→EC. Breast conservation is defined as tumorectomy, segmentectomy or quadrantectomy as a most radical surgery.
Toxicity of treatment | 24 weeks
  To assess the toxicity and compliance of PO→EC and to compare it with PCb→EC. Tolerability and safety will be assessed on the basis of adverse events, serious adverse events, adverse events of special interest and treatment discontinuations. Safety by toxicity grades is defined by the NCI-CTCAE version 4.0.

OTHER OUTCOMES:
Potential biomarkers predicting safety and compliance, like SNPs, TILs, PARP, 53BP1, REV7 and other biomarkers considered for breast cancer | 24 weeks
  To correlate co-occurring mutations detected by next generation sequencing in lymphocytes or in tumors cells with pCR (exploratory). Blood ampling before start of Treatment, after 12 and after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle 0 Loibl, Prof., MD, Study Chair — Sibylle Loibl, Prof., MD ASCO, ESGO, ESMO, DKG, DGGG, AGO, DGS, BIG, BCIRG, St. Gallen Faculty Member, SABCS Faculty member
Locations (12):
- Germany (12):
  - Kliniken Esslingen, Gynäkologie Onkologie, Esslingen am Neckar, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Onkologisches Zentrum am Rotkreuzklinikum München, München, Bavaria
  - Elisabeth Krankenhaus, Kassel, Hesse
  - Sana Klinikum Hameln-Pyrmont, Hamelin, Lower Saxony
  - Gemeinschaftspraxis, Hildesheim, Lower Saxony
  - Klinikum Südstadt, Rostock, Mecklenburg-Vorpommern
  - Marienhospital Witten, Witten, North Rhine-Westphalia
  - Martin-Luther-Universität Halle Wittenberg, Halle, Saxony-Anhalt
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal, Saxony-Anhalt
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - Praxisklinik, Berlin

REFERENCES:
- [Background] Von Minckwitz G, Timms K, Untch M, Elkin E P, Fasching P A, Schneeweiss A et al. Prediction of pathological complete response (pCR) by Homologous Recombination Deficiency (HRD) after carboplatin-containing neoadjuvant chemotherapy in patients with TNBC: Results from GeparSixto. J Clin Oncol 33, 2015 (suppl; abstr 1004)
- [Background] Tutt A, Ellis P, Kilburn L et al. The TNT trial: A randomized phase III trial of carboplatin (C) compared with docetaxel (D) for patients with metastatic or recurrent locally advanced triple negative or BRCA1/2 breast cancer. SABCS 2014.
- [Background] Sikov WM, Berry DA, Perou CM, Singh B, Cirrincione CT, Tolaney SM, Kuzma CS, Pluard TJ, Somlo G, Port ER, Golshan M, Bellon JR, Collyar D, Hahn OM, Carey LA, Hudis CA, Winer EP. Impact of the addition of carboplatin and/or bevacizumab to neoadjuvant once-per-week paclitaxel followed by dose-dense doxorubicin and cyclophosphamide on pathologic complete response rates in stage II to III triple-negative breast cancer: CALGB 40603 (Alliance). J Clin Oncol. 2015 Jan 1;33(1):13-21. doi: 10.1200/JCO.2014.57.0572. Epub 2014 Aug 4. PMID 25092775
- [Background] von Minckwitz G, Schneeweiss A, Loibl S, Salat C, Denkert C, Rezai M, Blohmer JU, Jackisch C, Paepke S, Gerber B, Zahm DM, Kummel S, Eidtmann H, Klare P, Huober J, Costa S, Tesch H, Hanusch C, Hilfrich J, Khandan F, Fasching PA, Sinn BV, Engels K, Mehta K, Nekljudova V, Untch M. Neoadjuvant carboplatin in patients with triple-negative and HER2-positive early breast cancer (GeparSixto; GBG 66): a randomised phase 2 trial. Lancet Oncol. 2014 Jun;15(7):747-56. doi: 10.1016/S1470-2045(14)70160-3. Epub 2014 Apr 30. PMID 24794243
- [Result] DOI: 10.1200/JCO.2019.37.15_suppl.506 Journal of Clinical Oncology 37, no. 15_suppl (May 20, 2019) 506-506. Fasching PA, Jackisch J, Rhiem K et al. GeparOLA: A randomized phase II trial to assess the efficacy of paclitaxel and olaparib in comparison to paclitaxel/carboplatin followed by epirubicin/cyclophosphamide as neoadjuvant chemotherapy in patients (pts) with HER2-negative early breast cancer (BC) and homologous recombination deficiency (HRD). J Clin Oncol 2019; 37.15_suppl.506; oral presentation
- [Derived] Fasching PA, Link T, Hauke J, Seither F, Jackisch C, Klare P, Schmatloch S, Hanusch C, Huober J, Stefek A, Seiler S, Schmitt WD, Uleer C, Doering G, Rhiem K, Schneeweiss A, Engels K, Denkert C, Schmutzler RK, Hahnen E, Untch M, Burchardi N, Blohmer JU, Loibl S; German Breast Group and Arbeitsgemeinschaft Gynakologische Onkologie Breast. Neoadjuvant paclitaxel/olaparib in comparison to paclitaxel/carboplatinum in patients with HER2-negative breast cancer and homologous recombination deficiency (GeparOLA study). Ann Oncol. 2021 Jan;32(1):49-57. doi: 10.1016/j.annonc.2020.10.471. Epub 2020 Oct 21. PMID 33098995
- See also: GeparOla website — http://www.gbg.de/de/studien/aktive-studien.php